CLINICAL TRIAL: NCT06937281
Title: A Phase II Trial Evaluating Stereotactic Ablative Radiotherapy for Primary and Regional Breast Tumors (SABR-PRIMeR)
Brief Title: SABR PRIMER - Evaluating Stereotactic Ablative Radiotherapy for Primary and Regional Breast Tumors
Acronym: SABR PRIMER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H25-00274
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Metastases
Keywords: SABR
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: A retrospective study will be conducted to create a matched cohort to compare locoregional control rates with patients who received conventional fractionated radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): SABR treatment to Whole breast +/- regional lymph nodes
  Interventions: Radiation: SABR

INTERVENTIONS:
Radiation: SABR — Prescription dose/fractionation: 26Gy/5 with 40Gy/5 +/- 35Gy/5 Boost Radiation Technique: VMAT Treatment Frequency: Every other day (EOD)

SUMMARY:
The study is being done to determine if stereotactic ablative radiotherapy (SABR) can control tumour growth for patients with metastatic breast cancer.

Secondary objectives will be overall survival, progression-free survival and time to switch of next line of systemic therapy.

Radiation-related adverse events will be assess, with a specific focus on dermatitis, lymphedema and brachial plexopathy.

The exploratory objective is to correlate toxicities and outcomes with peripheral blood biomarkers and circulating tumor DNA to potentially help predict responses in future patients receiving combined therapy.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to determine if stereotactic ablative radiotherapy (SABR) can provide effective locoregional control for patients with metastatic breast cancer. As secondary objectives, the investigators will assess the overall survival, progression-free survival and time to switch of next line of systemic therapy. The investigators will also assess radiation-related adverse events using CTCAE v5.0, with a specific focus on dermatitis, lymphedema and brachial plexopathy. Finally, as an exploratory objective, the investigators aim to correlate toxicities and outcomes with peripheral blood biomarkers and circulating tumor DNA to potentially help predict responses in future patients receiving combined therapy.

Primary Objective:

• Assess median, 1-year and 2-year locoregional control

Secondary Objectives:

* Assess median, 1-year and 2-year overall survival
* Assess median, 1-year and 2-year progression-free survival
* Assess median time to systemic therapy switch
* Assess radiation-related adverse events using CTCAE v5.0

Correlative Objectives:

• Correlate outcomes with peripheral blood-derived parameters

Research Design The trial is designed as a single-arm interventional study investigating stage IV breast cancer with persistent or progressive locoregional disease despite the use of standard systemic therapy A retrospective study will be conducted to create a matched cohort to compare locoregional control rates with patients who received conventional fractionated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed AJCC 7th/8th edition Stage IV invasive ductal carcinoma or invasive lobular carcinoma of the breast.
2. Measurable disease in the breast, suitable to receive radiotherapy.
3. Receiving or planned to receive systemic therapy.

   a. The following should be held for the duration of treatment: cytotoxic chemotherapy, CDK4/6 inhibitors, T-DXd
4. Patients are allowed to have SABR for oligometastatic disease as clinically indicated
5. Age 18 or older
6. ECOG Performance Status 0-2
7. Life expectancy greater than 6 months
8. Able and willing to provide informed consent
9. Able to complete patient reported outcome questionnaires

Exclusion Criteria:

1. Contraindications to radiotherapy, including a history of SLE, systemic scleroderma, IPF, ataxia telangiectasia, pregnancy
2. Previous history of locoregional radiotherapy to the ipsilateral breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Locoregional Control | 2 Years
  Assess median, 1-year and 2-year locoregional control

SECONDARY OUTCOMES:
Overall survival | 2 Years
  Assess median, 1-year and 2-year overall survival
Progression Free Survival | 2 Years
  Assess median, 1-year and 2-year progression-free survival
systemic therapy switch | 2 Years
  Assess median time to systemic therapy switch
Adverse Events | 2 Years
  Assess radiation-related adverse events using CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer - Vancouver, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided